CLINICAL TRIAL: NCT04726215
Title: Imaging of T-cell Activation With [18F]F-AraG in Advanced Non Small Cell Lung Cancer (NSCLC) Patients Undergoing PD-1/PD-L1 Directed Therapy
Brief Title: Imaging of T-cell Activation With [18F]F-AraG in Advanced Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CST-FARAG-IO-MULT-201
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: [18F]F AraG — PET imaging agent specific to activated T cells

SUMMARY:
This is a pilot study using [18F]F AraG PET imaging to evaluate the immunological response to checkpoint inhibitor therapy (CkIT) in patients with advanced NSCLC tumors at multiple study sites. The main objectives of the study are to quantify the change in [18F]F AraG PET signal before and after CkIT therapy, and to correlate this change in [18F]F AraG PET signal with a radiographic response.

DETAILED DESCRIPTION:
Approximately 50 patients will undergo two research PET/CT scans with [18F]F AraG at two time points. Each patient will receive two 5 (+/-10%) mCi doses of [18F]F AraG, one for each imaging time point. Eligible subjects will undergo a pre-treatment [18F]F AraG PET/CT scan within 7 days prior to treatment, followed by treatment, and an on-treatment [18F]F AraG PET/CT within 7-14 days of treatment.

Objectives:

* Quantify [18F]F-AraG uptake in advanced NSCLC tumor (primary, nodal, and metastatic sites) at baseline and after 1 dose of anti-PD-1/PD-L1 therapy in patients treated with standard of care immunotherapy (as monotherapy or part of combination therapy).
* Correlate change in [18F]F AraG uptake in tumor lesions with radiographic response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically confirmed NSCLC and planned to undergo immunotherapy as monotherapy or as combination therapy with concurrent as treatment for advanced/metastatic disease.
2. RECIST measurable disease.
3. ECOG performance status of 0, 1 or 2.
4. Life expectancy >/= 6 months at enrollment.

Exclusion Criteria:

1. Serious comorbidities that in the opinion of the investigator/sponsor could compromise protocol objectives.
2. Pregnant women or nursing mothers.
3. Patients with severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
[18F]F-AraG uptake signal | two years
  [18F]F-AraG uptake signal will be measured quantitatively by SUV-bw of the tumor volumes of interest before and after undergoing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Behera, MD, Principal Investigator — CellSight Technologies, Inc.
Locations (3):
- United States (3):
  - Palo Alto Veterans Institute of Research, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Stony Brook University, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No